CLINICAL TRIAL: NCT07266454
Title: Evaluating Stumble Recovery Functions of Prosthetic Knees
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CIP2025012117
Record Dates: First submitted 2025-09-02; First posted 2025-12-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fall Prevention; Balance, Falls; Amputation of Lower Limb
Keywords: amputation; falls; fall prevention; balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comprehensive Evaluation of Prosthetic Knee Devices (Experimental): Participants enrolled in this protocol will take part in one or more sequential study phases, including formative evaluation, verification, validation, and/or comparative crossover assessment. Depending on study design and eligibility, participants may contribute to different phases, such as providing feedback on iterative prototypes (formative phase), verifying device functions (verification phase), validating device effectiveness and safety in simulated real-world conditions (validation phase), or participating in randomized crossover comparisons of device performance with various configurations and/or comparator devices (comparative phase). Each participant will be exposed to the relevant device configurations and study conditions for the specific phase(s) in which they are enrolled.
  Interventions: Device: Prosthetic Knee (e.g Power Knee, Navii, Rheo Knee, ...)

INTERVENTIONS:
Device: Prosthetic Knee (e.g Power Knee, Navii, Rheo Knee, ...) — Participants will use one or more investigational prosthetic knee devices, which may include [list trade names, e.g., Navii, Rheo Knee, Power Knee], under different conditions as part of one or more study phases, including formative evaluation, verification, validation, and/or comparative crossover assessment. The study may include multiple device configurations or models within the prosthetic knee class, and comparative assessment against standard of care or alternative prosthetic knee devices as applicable.

SUMMARY:
The study aims to conduct a formative evaluation, along with verification, validation, and comparative analysis of the stumble recovery function in prosthetic devices by collecting relevant clinical data. The study will involve participants who are current users of lower-limb prosthetics. Utilizing a robust study design, data will be gathered in both controlled setting and real-world to thoroughly assess the performance, safety, and user satisfaction of the function. The scientific value of this research lies in its potential to enhance prosthetic technology, support evidence-based clinical practices, and ultimately improve the quality of life for users by reducing fall risks and increasing mobility confidence.

ELIGIBILITY:
Inclusion Criteria:

* 40 kg < body weight < 136kg
* Cognitive ability to understand all instructions and questionnaires in the study
* Willing and able to participate in the study and following the protocol
* Age ≥ 18 years
* Able to walk independently without the use of assistive device such as a cane or walker
* Regular prosthesis users for at least 1 year with unilateral lower limb amputation at or below the transfemoral level (or equivalent level limb deficiency)

Exclusion Criteria:

* Users with pain which can affect their mobility
* Users with socket comfort score less than 7
* Users with cognitive impairment
* Pregnant Users
* Musculoskeletal disorders or neurological conditions that affect motor function, gait or balance
* Use of medications that are known to impair balance and coordination
* Any other conditions deemed by the investigator to make participation unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
User-Perceived Safety During Use of Stumble Recovery Function Assessed by 3-Point Scale | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  Safety perception will be assessed using a study-specific 3-point scale. Participants will rate their perception of safety when using the investigational device with the stumble recovery function enabled, compared to either a previous device version without this function or other similar devices. For each aspect of the new function, users will report a score: worse (0), neutral (1), or better (2).
Expert-Perceived Safety of Stumble Recovery Assessed by 3-Point Scale | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  Safety perception will be assessed by researchers or engineers using a study-specific 3-point scale. Experts will rate the safety of the investigational device with the stumble recovery function enabled, compared to either a previous device version without this function or other similar devices. For each aspect of the new function, experts will report a score: worse (0), neutral (1), or better (2)
User-Perceived Stability and Confidence | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  Stability and confidence rated by users (worse/neutral/better) via observation and feedback after using the new function.
Fall Rate Following Induced Perturbation Events Assessed by Direct Observation | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  The outcome will be measured as the fall rate following induced perturbation events during use of the stumble recovery function. The fall rate is defined as the number of perturbation events resulting in falls divided by the total number of perturbation events, assessed by direct observation and/or video recording during controlled laboratory testing. The reduction in fall rate will be compared to baseline conditions, which may include use of non-microprocessor-controlled knees (NMPKs) or microprocessor-controlled knees (MPKs) without the stumble recovery function.
Stumble and Fall Detection Rate Assessed by Device Log Analysis | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  The detection rate will be measured as the proportion of induced stumbles and falls (during controlled perturbation events) that are automatically identified by the knee's stumble recovery system. Detection will be confirmed via analysis of device event logs, which record when the system recognizes a stumble or fall. The successful detection rate is defined as the number of correctly detected stumbles and falls divided by the total number of perturbation events.
Stumble and Fall Response Trigger Rate Assessed by Device Log Analysis | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  The response trigger rate will be measured as the proportion of detected stumbles and falls that result in the knee successfully initiating the appropriate response, as confirmed by device event logs. For each instance where a stumble or fall is detected by the knee's system, device logs will be analyzed to verify whether the corresponding response (e.g., stumble recovery activation, fall dampening) was triggered. The trigger rate is defined as the number of successful response triggers divided by the total number of detected stumbles and falls.
Stumble and Fall False Detection Rate Assessed by Device Log Analysis | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  The false detection rate will be measured as the proportion of incorrectly detected stumbles or falls by the knee's system, as determined through analysis of device event logs during controlled testing sessions. A false detection is defined as a device-logged stumble or fall event that does not correspond to an actual perturbation or loss of balance observed by study personnel. The false detection rate is calculated as the number of incorrect detections divided by the total number of detections of stumbles and falls.
Stumble Recovery False Trigger Rate Assessed by Device Log Analysis Stumble Recovery False Trigger Rate Stumble Recovery False Trigger Rate | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  The false trigger rate will be measured as the proportion of incorrect activations of the knee's stumble recovery function, determined by analysis of device event logs during controlled testing sessions. A false trigger is defined as activation of the stumble recovery response by the device in the absence of a true stumble or fall event, as verified by study personnel or video review. The false trigger rate is calculated as the number of incorrect triggers divided by the total number of stumble recovery activations.
  Measures how often the knee's stumble recovery is incorrectly activated during testing.
Fear of Falling Reduction Assessed by Falls Efficacy Scale-International (FES-I) | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  Changes in fear of falling will be assessed using the Falls Efficacy Scale-International (FES-I) questionnaire. The FES-I provides a total score representing the participant's concern about falling during social and physical activities. Scores range from 16 (no concern about falling) to 64 (severe concern about falling); higher scores indicate a greater fear of falling. The outcome will be measured as the change in FES-I score from baseline (prior to use of the stumble recovery function) to after using the device with the stumble recovery function enabled.
Perceived Safety and Balance Assessed by Activities-specific Balance Confidence (ABC) Scale | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  Perceived safety and balance will be assessed using the Activities-specific Balance Confidence (ABC) Scale questionnaire. The ABC Scale measures an individual's confidence in maintaining balance during various daily activities. Scores range from 0% (no confidence) to 100% (complete confidence); higher scores indicate better perceived safety and balance. The outcome will be measured as the change in ABC Scale score from baseline (using the prescribed or previous knee) to after using the device with the stumble recovery function enabled. Non-inferiority will be established if the change in score is within the minimal detectable change (MDC), set at 11.56 percentage points.
Stumble Recovery Ability Assessed by Motion Capture or Wearable Sensor Analysis | Assessed at the end of each device exposure period within formative (1 day use), verification (1 day use), validation (1 day use), and crossover phases (1-3 weeks use per exposure), at scheduled visits.
  Improvement in stumble recovery ability will be assessed by measuring recovery time, defined as the duration from stumble onset to regaining stable posture. Recovery time will be recorded during controlled perturbation events using motion capture technology or wearable sensors. Shorter recovery times indicate enhanced ability to recover from stumbles with the stumble recovery function enabled, compared to baseline device conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Thor Fridriksson, Doctor, Principal Investigator — Össur Iceland ehf
Locations (2):
- Iceland (2):
  - University of Iceland, Reykjavik
  - Össur Iceland ehf., Reykjavik

IPD SHARING:
Plan to Share IPD: No